CLINICAL TRIAL: NCT01770717
Title: Assessment of the Potential for Pressure Ulcer Formation Using a New Optical Imaging Technology: Spatial Frequency Domain Imaging
Brief Title: Assessment of the Potential for Pressure Ulcer Formation
Status: Withdrawn | Type: Observational
Why Stopped: Not NIH defined clinical trial study.
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Anthony Durkin, Ph.D. Associate Professor, Director, Laboratory for Functional Imaging and Spectroscopy of Superficial Tissues, University of California, Irvine
Other Study IDs: 20128868
Record Dates: First submitted 2013-01-14; First posted 2013-01-18 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Pressure Ulcer Not Visible

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pressure Ulcer Formation: Assessment of Pressure Ulcer Formation using Spatial Frequency Domain Imaging
  Interventions: Other: Spatial Frequency Domain Imaging

INTERVENTIONS:
Other: Spatial Frequency Domain Imaging — Assessment of Pressure Ulcer Formation using Spatial Frequency Domain Imaging

SUMMARY:
Pressure ulcers are a significant problem in institutionalized, elderly, and critically ill patients. Pressure ulcers result in significant pain, changing quality of life, and often leading to significant morbidity and prolonged hospital stays, and ultimately increased the healthcare cost.

According to the International Pressure Ulcer Prevalence Survey, the prevalence of hospital acquired pressure ulcers in the United States was 13.5% in 2008 and 12.8% in 2009. This survey also indicated that the highest rate of pressure ulcers is in the long term acute care population (22%).

DETAILED DESCRIPTION:
Researchers developed a non-contact optical imaging technology call Spatial Frequency Domain Imaging which can identify the tissue regions that are at risk of developing pressure ulcers prior to development of irreversible tissue damage. The Spatial Frequency Domain Imaging can identify metabolic and biochemical differences in the tissues near bony prominences which are at risk for developing pressure ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age and older
* Diagnose with potential of pressure ulcers

Exclusion Criteria:

* No potential of pressure ulcers
* Has history of vascular disease in both lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study polpulation will be selected from UCIMC Inpatient care unit
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Formation of Pressure Ulcer | up to 6 months
  Assessment of Pressure Ulcer Formation using Spatial Frequency Domain Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Durkin, PhD, Principal Investigator — Beckman Laser Institute, UCI
Locations (1):
- UCIMC, Orange, California, United States